CLINICAL TRIAL: NCT00538889
Title: Combined Administration of Lecozotan SR and Citalopram: a Double Blind, Multiple Dose Study in Young Healthy Subjects
Brief Title: Study Evaluating a Combined Administration of Lecozotan SR and Citalopram in Young Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3098B1-134
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
Keywords: Adult
MeSH Terms: interventions — lecozotan; Citalopram

INTERVENTIONS:
Drug: Lecozotan SR
Drug: Citalopram

SUMMARY:
To assess the safety and tolerability of lecozotan SR and citalopram when coadministred to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated IRB/IEC-approved informed consent form before any study-specific screening procedures are performed.
* Men or women aged 18 to 50 years, inclusive, at screening.
* Women of nonchildbearing potential, defined as being surgically sterile or postmenopausal for > 1 year, may be included. For women below 50 years of age, at least two years of retrospective amenorrhea and FSH>38 and estrogen <20 are required.
* Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight greater than or equal to 50 kg. BMI is calculated by taking the subject's weight, in kilograms, divided by the square of the subject's average height, in meters, at screening: BMI = weight (kg)/(height [m])2

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any clinically important deviation from normal limits in physical examination, vital signs, 12-lead ECGs, or clinical laboratory test results.
* Hypersensitivity to citalopram or any of the inactive ingredients in citalopram.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of 5-HT toxicity (Hunter serotonin toxicity criteria) and CNS questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Manchester, United Kingdom